CLINICAL TRIAL: NCT07001891
Title: Functional Connectivity of the Interoceptive Network in Restless Legs Syndrome (RLS) : an Anatomical-clinical Prospective Study Based on Daily-life Assessment
Brief Title: Functional Connectivity of the Interoceptive Network in RLS
Acronym: IntoRLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Restless Legs Syndrome Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/68
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; Interoception; Insular Cortex; Functional Connectivity
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restless Legs Syndrome (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: auto-questionnaires (PSQI, ISI, ESS and HADS); Device: Ecological Momentary Assessment (EMA); Device: activity-rest cycle; Behavioral: auto-questionnaires (ASRS, PSAS, APS, MAIA-2); Device: MRI
- healthy controls (Active Comparator)
  Interventions: Behavioral: auto-questionnaires (PSQI, ISI, ESS and HADS); Device: Ecological Momentary Assessment (EMA); Device: activity-rest cycle; Behavioral: auto-questionnaires (ASRS, PSAS, APS, MAIA-2); Device: MRI

INTERVENTIONS:
Other: Clinical assessment — RLS history, RLS treatments, and International Restless Legs Syndrome Rating Scale (IRLSRS) will be recorded
  Arms: Restless Legs Syndrome
Behavioral: auto-questionnaires (PSQI, ISI, ESS and HADS) — To evaluate sleep quality, daytime somnolence and mood disorders (Pittsburgh Sleep Quality Index (PSQI), Insomnia Severity Index (ISI), Epworth Sleepiness Scale (ESS) and Hospital Anxiety and Depression Scale (HADS)).
Device: Ecological Momentary Assessment (EMA) — 4 electronic interviews administered per day during 14 days by a study-dedicated Android OS smartphone
Device: activity-rest cycle — To further investigate the mutual influence of sleep quality on RLS symptoms and mood, the activity-rest cycle will be monitored by wearable actigraph to be placed on the non-dominant wrist during a period of 13 days and 14 nights.
Behavioral: auto-questionnaires (ASRS, PSAS, APS, MAIA-2) — Interoceptive awareness and accuracy estimation : Adult ADHD Self-Report Scale (ASRS), Pre-Sleep Arousal Scale (PSAS), Arousal Predisposition Scale (APS) et Multidimensional Assessment of Interoceptive Awareness version 2 (MAIA-2)
Device: MRI — Morning and evening functional brain imaging

SUMMARY:
Restless Legs Syndrome (RLS) is a sensorimotor disorder primarily characterized by an irresistible urge to move the legs while at rest. A key hypothesis suggests that RLS symptoms are linked to abnormal brain function in processing internally generated stimuli, particularly interoception. This distorted perception of the internal bodily state leads to maladaptive behaviors, which may manifest across a wide range of medical and psychiatric disorders. Here, the investigators hypothesize that dysfunction in the insular cortex (IC) may result in a failure of behavioral adaptation, primarily expressed as an urge to move the legs and hyperarousal, even when the body and mind need rest. This project aims to assess the relationship between interoceptive abilities and diurnal fluctuations in IC functional connectivity (FC) in patients with RLS compared to healthy controls. The investigators will also examine correlations between the FC of the interoceptive network, measured in the morning and evening on the same day, using multilayer network analysis, daily fluctuations in RLS symptom severity, and objective measurements of the sleep/wake cycle, gathered through a two-week ambulatory assessment using mobile technologies such as Ecological Momentary Assessment (EMA) and actigraphy, along with scores from self-reported questionnaires. The findings may provide strong evidence to support or refute the hypothesis of interoceptive dysfunction in RLS patients.

DETAILED DESCRIPTION:
Despite extensive research into the pathophysiology of RLS, no unified mechanism has been identified to explain the prominent clinical features of the disorder, including both sensorimotor and non-motor symptoms. One plausible hypothesis is that RLS symptoms are related to abnormal brain function in processing internally generated stimuli, particularly interoception. Distorted perceptions of the internal bodily state can lead to maladaptive behaviors, which may manifest in a wide range of medical disorders, including RLS, attention-deficit/hyperactivity disorder (ADHD), insomnia, eating disorders/obesity, fibromyalgia, and psychiatric conditions. The interoceptive abilities of RLS patients, specifically their capacity to perceive and assess their internal bodily state, have not been extensively studied, despite their potential to deepen our understanding of the sensorimotor discomfort in the legs and associated non-motor symptoms. The IntoRLS project will therefore precisely characterize the temporal variation in symptom severity and interoceptive awareness in RLS patients, alongside their sleep/wake cycle disturbances, using ambulatory assessments. This ecological assessment will be linked to time-of-day variations in intrinsic insular connectivity, assessed via functional brain imaging. At the inclusion visit, eligible participants (both patients and matched controls) will be provided with a study-dedicated smartphone for a two-week period, as well as a wearable actigraph to monitor their activity/rest cycles. Participants will complete self-reported questionnaires assessing the severity of RLS symptoms, ADHD symptoms, anxiety and depression, daytime sleepiness, and arousal predisposition. At the end of the participation period (J+14), participants will undergo functional brain imaging sessions in the morning and evening. Between the two sessions, each participant will complete the Multidimensional Assessment of Interoceptive Awareness (MAIA-2) questionnaire and perform the Heartbeat Detection Task to evaluate interoceptive accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Person aged from 18 to 70 years
* Only for the patients : ny patient with a diagnosis of idiopathic RLS based on medical history and the presence of the 5 RLS diagnostic criteria
* Normal clinical examination
* Person affiliated or benefiting from a social security scheme
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and prior to any review required by the research).

Exclusion Criteria:

* Any significant psychiatric illness or mood disorder
* History or presence of chronic pain other than that associated with RLS, history of epilepsy or serious head injury, history of peripheral neuropathy, diabetes
* Clinically significant sleep apnea, narcolepsy, or any secondary causes of RLS (e.g. chronic renal failure/hemodialysis, pregnancy)
* Other active clinically significant illness, including unstable cardiovascular, or neoplasic pathology which could interfere with the study conduct or interfere with study assessments or compromise the study participation
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia or refusing MRI)
* Pregnant or breastfeeding woman
* Persons referred to in articles L.1121-5 to L.1121-8 (persons deprived of liberty by judicial or administrative decision, minors, adults subject to a legal protection measure or unable to express their consent).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity (FC) of the anterior and posterior insular cortex (IC) measured at rest. | 14 days after baseline (Day 0)
  The investigators hypothesize that this connectivity will differ between patients and control subjects.
  This outcome will be assessed through the temporal fluctuation of the BOLD signal measured during the MRI examination conducted in the morning and again in the evening.

SECONDARY OUTCOMES:
Correlations will be explored between the scores obtained by patients and those of the healthy volunteer group on the various self-assessment scales. | 14 days after baseline (Day 0)
  Score comparisons on these same scales will also be conducted between the patient group and the healthy volunteer group. The scores analyzed will be those obtained on the following scales:
  * International Restless Legs Syndrome Rating Scale (IRLSRS) (to assess the severity of RLS),
  * Insomnia Severity Index (ISI),
  * Adult ADHD Self-Report Scale (ASRS) (to screen for symptoms of ADHD),
  * Hospital Anxiety and Depression Scale (HADS) (to assess levels of depression and anxiety),
  * Multidimensional Assessment of Interoceptive Awareness Version 2 (MAIA-2) (to evaluate interoceptive awareness),
  * Pre-Sleep Arousal Scale (PSAS) and Arousal Predisposition Scale (APS) (to measure levels of hypervigilance),
  * Epworth Sleepiness Scale (ESS) (to assess hypersomnolence).
Correlations will be explored between the severity score of the RLS and sleep parameters | 14 days after baseline (Day 0)
  assessed by actigraphy (specific measures including: Total Sleep Duration [minutes], Sleep Efficiency [%], Wake After Sleep Onset [minutes], and Sleep Onset Latency [minutes]) as well as scores from Ecological Momentary Assessment smartphone questionnaires.
Correlations will be explored between altered functional connectivity of the patients' insular cortex | 14 days after baseline (Day 0)
  (measured by statistical synchrony or temporal correlation of BOLD [Blood Oxygen Level Dependent] signals across different brain regions) and sleep parameters assessed by actigraphy (specific measures including Total Sleep Duration [minutes], Sleep Efficiency [%], Wake After Sleep Onset [minutes], and Sleep Onset Latency [minutes]) as well as scores from Ecological Momentary Assessment smartphone questionnaires.
  Comparisons will also be made with results obtained from the healthy volunteer group.

CONTACTS AND LOCATIONS:
Overall Officials: Imad Marc Antoine GHORAYEB, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Gwénaëlle CATHELINE, PhD, Study Chair — Université de Bordeaux - INCIA
Locations (1):
- CHU de Bordeaux - Neurophysiologie Clinique de l'Enfant et de l'Adulte, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No